# Informed consent

Detection of Clinical-functional Changes Following Exercise Therapy and Education in Institutionalised and Community-dwelling Older Adults Diagnosed with Sarcopenia

N°: 101//2022

## MODELO DE CONSENTIMIENTO INFORMADO

PROYECTO: Detection of Clinical-functional Changes Following Exercise Therapy and Education in Institutionalised and Community-dwelling Older Adults Diagnosed with Sarcopenia

Sujeto muestral ID#:

Centro: FACULTAD DE MEDICINA Y CIENCIAS DE LA SALUD Centro ID#: UNIVERSIDAD DE

**EXTREMADURA** 

**Investigador: LUIS ESPEJO ANTÚNEZ** 

LEA DETENIDAMENTE LA INFORMACIÓN CONTENIDA EN ESTE DOCUMENTO Y ASEGÚRESE QUE ENTIENDE ESTE PROYECTO DE INVESTIGACIÓN. POR FAVOR SI ESTA DE ACUERDO EN PARTICIPAR EN ESTE ESTUDIO, FIRME ESTE DOCUMENTO. POR SU FIRMA RECONOCE QUE HA SIDO INFORMADO DE LAS CARACTERÍSTICAS DEL PROYECTO, DE SUS REQUISITOS Y SUS RIESGOS Y QUE ACEPTA LIBREMENTE PARTICIPAR EN ÉL. UNA COPIA DEL PRESENTE DOCUMENTO LE SERÁ ENTREGADA.

## OBJETO DEL ESTUDIO.

Participar como sujeto muestral en un estudio de investigación experimental, de carácter prospectivo, dirigido a conocer los efectos derivados de una intervención mediante ejercicio terapéutico o su combinación con estimulación eléctrica neuromuscular.

## PROCEDIMIENTOS Y DURACIÓN DEL ESTUDIO.

El procedimiento al que será sometido/a será:

- VALORACIÓN INICIAL DE PARÁMETROS CLÍNICO-FUNCIONALES
- INTERVENCIÓN MEDIANTE UN PROGRAMA DE EJERCICIO TERAPÉUTICO DE FUERZA DURANTE 12 SEMANAS (2 VECES SEMANA), CON UNA DURACIÓN APROXIMADA DE 45 MINUTOS.
- VALORACIÓN FINAL Y SEGUIMIENTO TRAS LA FINALIZACIÓN DEL PROGRAMA

Los datos obtenidos serán utilizados exclusivamente con finalidad de investigación sin ánimo de lucro.

## RESULTADOS DEL ESTUDIO.

Al finalizar el estudio se le informará del resultado global del mismo si usted lo desea, pero NO de su resultado personal, que se tratará con total confidencialidad de acuerdo con la Declaración de Helsinki y la Ley 14/2007, de Investigación biomédica.

## RIESGOS DERIVADOS DE LA PARTICIPACIÓN EN EL ESTUDIO.

-. LOS RIESGOS ASOCIADOS A LA PARTICIPACIÓN EN EL ESTUDIO SE CIRCUNSCRIBEN A LOS CRITERIOS DE EXCLUSIÓN INDICADOS ANTES DEL INICIO DEL ESTUDIO. DE MANERA POCO HABITUAL, EL SUJETO QUE RECIBE ESTIMULACIÓN ELÉCTRICA DENTRO DEL PROGRAMA DE

EJERCICIO TERAPÉUTICO DE FUERZA PUEDE PRESENTAR ALGÚN INDICIO DE APRENSIÓN PSICOLÓGICA (AVERSIÓN A LA CORRIENTE ELÉCTRICA CON PUNTUACIONES INFERIORES A 45 PUNTOS EN ESCALA DE APRENSIÓN PSICOLÓGICA PERSONAL) Y FATIGA MUSCULAR TRAS EJECUTAR LA INTERVENCIÓN.

#### BENEFICIOS.

La participación en el proyecto no será recompensada económicamente. Aparte de lo comentado anteriormente, se estima que el desarrollo del estudio en el que participará aportará beneficios relevantes en lo que a la mejora del conocimiento respecta sobre intervenciones fisioterapéuticas para la prevención y mejora de la sarcopenia en el adulto mayor.

## COSTES.

Su participación no le supondrá ningún coste.

El investigador principal LUIS ESPEJO ANTÚNEZ, puede ser contactado en cualquier momento en el siguiente teléfono 650057024 a fin de recabar información acerca del proyecto y en la siguiente dirección:

Departamento de Terapéutica Médico-quirúrgica Facultad de Medicina Av. de Elvas 06071Badajoz

## CONFIDENCIALIDAD

De acuerdo con la normativa legal vigente, los resultados del estudio se tratarán con total confidencialidad. El protocolo de recogida de datos será archivado, y a cada participante se le asignará una clave de tal modo que no pueda relacionarse la información obtenida con la identidad del sujeto

El investigador principal del proyecto se compromete a que la confidencialidad de los datos que se puedan obtener en dicho proyecto será escrupulosamente observada, y que los datos personales de los sujetos participantes no serán conocidos por los investigadores del proyecto. En los casos que corresponda, éstos informarán al responsable médico o a los afectados si creen que algún resultado del proyecto podría ser de su interés.

El investigador principal del proyecto se compromete a no utilizar los resultados para otros estudios diferentes a los de este proyecto y a no traspasar los resultados a otros posibles proyectos o equipos de investigación.

Para todo lo no previsto en este documento, se aplicará la legislación vigente sobre protección de datos de carácter personal (Ley 41/2002, de 14 de noviembre, básica reguladora de la autonomía del paciente y de derechos y obligaciones en materia de información y documentación clínica, BOE 274 de 15 de noviembre de 2002; Ley Orgánica 15/1999, de 13 de diciembre, de Protección de Datos de Carácter Personal; BOE 298 de 14 de diciembre de 1999; Real Decreto 1720/2007, de 21 de diciembre, por el que se aprueba el Reglamento de desarrollo de la Ley Orgánica 15/1999, de 13 de diciembre, de protección de datos de carácter personal, BOE 17 de 19 de enero de 2008), sobre investigación biomédica (Ley 14/2007, de 3 de julio, de Investigación biomédica; BOE 159 de 4 de julio de 2007) y cualquier otra que resultara aplicable.

Los resultados del estudio pueden ser publicados en revistas científicas o publicaciones de carácter general. No obstante, la información concerniente a su participación será mantenida como confidencial.

Recibirá una copia de esta hoja de información y del consentimiento informado firmado por usted.

## DECLARACIÓN DEL PARTICIPANTE.

He sido informado por el personal relacionado con el proyecto mencionado:

- De las ventajas e inconvenientes, de la finalidad del estudio así como que mis resultados serán proporcionados de forma anónima a los investigadores del proyecto.
- Que he comprendido la información recibida y he podido formular todas las preguntas que he creído oportunas.

| Usted tiene derecho de participar o no en la invest | igación y de retirar su consentimiento en cualquie |
|---|---|
| momento. | |
| SE ME HA PROPORCIONADO COPIA DEL PRESENTE DOCUME | NTO. |
| Nombre: | Firma: |
| Declaración del profesional que ha informado | debidamente al participante. |
| Nombre: LUIS ESPEJO ANTÚNEZ | Firma: |